CLINICAL TRIAL: NCT00286806
Title: An Open-Label, Multicenter, Phase I/II Study of Single-Agent AT-101 in Men With Hormone Refractory Prostate Cancer (HRPC) and Rising Prostate Specific Antigen (PSA) Levels Who Have Not Received Prior Chemotherapy
Brief Title: A Study of Single-Agent AT-101 in Men With Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ascenta Therapeutics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-101-CS-006
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Hormone Refractory Prostate Cancer
MeSH Terms: interventions — gossypol acetic acid

INTERVENTIONS:
Drug: AT-101

SUMMARY:
This is an open-label, multicenter Phase I/II study to evaluate the safety and efficacy of single-agent AT-101 in men with hormone-refractory prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Rising PSA, as defined by increasing levels on at least two consecutive assessments
2. ECOG performance status 0 or 1
3. Adequate hematologic function
4. Adequate liver and renal function
5. Able to swallow and retain oral medication.

Exclusion Criteria:

1. Received prior chemotherapy for HRPC.
2. Concurrent therapy for the treatment of prostate cancer.
3. Clinical signs or symptoms of CNS metastases
4. Requirement for corticosteroid treatment, with the exception of topical corticosteroids or inhaled corticosteroids for reactive airway disease.
5. Active secondary malignancy or history of other malignancy within the last 5 years.
6. Failure to recover from toxicities related to prior therapy.
7. Uncontrolled concurrent illness.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27
Dates: Start 2005-12; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events.

SECONDARY OUTCOMES:
Complete or partial remission of disease

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, MD, Study Director — Ascenta Therapeutics, Inc.
Locations (4):
- United States (4):
  - Greenbrae, California
  - New Haven, Connecticut
  - Memphis, Tennessee
  - Madison, Wisconsin